CLINICAL TRIAL: NCT04952155
Title: A Single-center, Open-label Clinical Study to Evaluate the Efficacy and Safety of Low-dose IL-2 in the Treatment of Immune-associated ALS Syndrome
Brief Title: Low Dose IL-2 in the Treatment of Immune-associated ALS Syndrome
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: M2020420
Record Dates: First submitted 2021-06-27; First posted 2021-07-07 (Actual); Last update posted 2021-08-18 (Actual); Status verified 2021-06

CONDITIONS: Amyotrophic Lateral Sclerosis
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis | interventions — Interleukin-2

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- IL-2 (Experimental): The administration period was divided into 6 courses. 6 cycles of IL-2 were administered subcutaneously at a dose of 1 million IU every other day for 2 weeks, followed by a 2-week break in treatment.
  Interventions: Drug: IL-2

INTERVENTIONS:
Drug: IL-2 — The administration period was divided into 6 courses. 6 cycles of IL-2 were administered subcutaneously at a dose of 1 million IU every other day for 2 weeks, followed by a 2-week break in treatment. The adminstration course was 24 weeks.. The 24-week follow-up period was followed after the treatment.

SUMMARY:
The purpose of this study was to evaluate the efficacy and safety of low-dose IL-2 in the treatment of immunorelated ALS syndrome.

DETAILED DESCRIPTION:
This is a single-center, open-label, self-controlled clinical study with a sample size of 10 patients for 48 weeks, including 24 weeks of administration, and 24 weeks of follow-up. During the administration period, medication was given for 2 weeks and rest for 2 weeks, as a course of treatment, with a total of 6 courses for 24 weeks. During the administration period, the drug was given on alternate days, and IL-2 1mIU was subcutaneously injected the next day for 7 times, and then rested for 2 weeks, and the cycle was repeated for 6 times. The primary outcome index was the change in the rate of ALSFRS-R score between administration period and follow-up period. Secondary outcome measures included changes in the rate of ALSAQ-40 score, ROADS score, MRC score, survival time, FVC%, Treg and CD4+ T cell subsets, inflammatory factors, serum and cerebrospinal fluid NFL during follow-up versus administration , changes in the inhibition function of Treg; Exploratory outcome indicators included the change degree of compound muscle action potential (CMAP) amplitude, quantitative analysis of corneal nerve morphologic changes by corneal confocal microscopy (CCM), Treg single-cell sequencing transcriptome analysis. The related safety indexes were also evaluated.

ELIGIBILITY:
Inclusion Criteria:

* 18-70 years old;
* Clinically diagnosed with ALS syndrome, i.e., with ALS -like manifestations, consisting of a combination of upper and/or lower motor neuron damage;
* significant abnormalities with rheumatoid immune-related indicators, or diagnoses of immune-mediated ALS syndrome, including but not limited to multifocal motor neuropathy (MMN), Lewis-Sumner syndrome, and other ALS-like syndromes with an immune background that cannot be clearly classified;
* Poor treatment with conventional hormones or gamma globulin;
* Permitted concomitant treatment: oral prednisone or equivalent doses of other glucocorticoids (≤1.0mg/kg/d); Oral routine dose of immunosuppressants or immunomodulators, such as cyclophosphamide, tacrolimus, etc.; Routine oral doses such as too much force; Doses and types of accompanying therapeutic drugs should not be changed from the trial enrollment to the end of follow-up.
* For women of reproductive age, contraception for at least 2 weeks at the time of enrolment and negative urine HCG;
* Reasonable and effective contraceptive measures should be taken by subjects of childbearing age from the time of trial enrollment to the end of follow-up;
* Signed informed consent.

Exclusion Criteria:

* Allergic or intolerance to IL2;
* Receive non-standard treatment or use of excessive dose of glucocorticoids or gamma globulin intravenously within 2 months before enrollment;
* Vaccination within 6 months before enrolment or between enrolment and the end of follow-up;
* Peripheral venous white blood cells < 2000/mm3, lymphocytes < 600/mm3, platelets < 80,000 /mm3;
* Complicated with severe infection or inflammation, such as bacteremia, sepsis, etc.;
* Complicated blood system diseases, infectious diseases (hepatitis, HIV, tuberculosis, etc.), mental diseases, dementia, severe hypotension, substance abuse history, malignant tumor history, organ transplantation history, etc.;
* Severe liver, kidney, lung or heart dysfunction: heart failure (≥NYHA grade III), renal insufficiency (creatinine clearance ≤30ml/min), abnormal liver function (3 times the upper limit of normal >);
* Pregnant and lactating women;
* Currently participating in other clinical studies or using other investigational drugs.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Estimated)
Dates: Start 2020-01-01 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
ALSFRS-R score | week 0，week 24 and week 48
  Changes in the rate of ALSFRS-R score during administration period compared with follow-up period

SECONDARY OUTCOMES:
ALSFRS-R score | week 0，week 24 and week 48
  Changes in the slope of ALSFRS-R score during adminstration period compared with the follow-up period
ROADS score | week 0，week 24 and week 48
  Changes in the rate of ROADS score during adminstration period compared with the follow-up period
ALSAQ-40 score | week 0，week 24 and week 48
  Changes in the rate of ALSAQ-40 score during adminstration period compared with the follow-up period
MRC score | week 0，week 24 and week 48
  Changes in the rate of ALSAQ-40 score during adminstration period compared with the follow-up period
Immunological Responses | week 0 and week 24
  Analysis regulatory CD4+ T (Treg) cells , interleukin 17 (IL-17)-producing helper T (Th17) cells，Teff cells，follicular helper T (Tfh) cells and related cytokines before and during IL-2 treatment.
NFL in the serum and cerebrospinal fluid | week 0，week 24 and week 48

CONTACTS AND LOCATIONS:
Overall Officials: Dongsheng Fan, Principal Investigator — Peking University Third Hospital
Locations (1):
- Peking University Third Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Yes